CLINICAL TRIAL: NCT01733927
Title: An Evaluation of an Oral Rapid Test for HIV
Brief Title: An Evaluation of a Rapid Test for HIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: DIEECII #3
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: HIV Seropositivity
Keywords: HIV screening; Rapid test for HIV
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rapid testing for HIV (Experimental): The intervention consisted in administer an oral rapid test for HIV (OQA) to people that also had taken an ELISA test to compare their tests results. Group 1 consisted of 344 participants who did not know their HIV status; Group 2 consisted of 153 participants who were previously confirmed to be HIV positive. The participants were instructed to obtain their own oral fluid sample using the testing devices provide by the OQA rapid test kits. Project team members, certified to interpret OQA results, registered each test outcome on a data form using the same code number that the participant was assigned for the ELISA test.
  Interventions: Device: Rapid testing for HIV

INTERVENTIONS:
Device: Rapid testing for HIV — The research team members were trained and certified in administering the OQA testing through the AIDS International Consortium in Philadelphia (WHCI), USA. During the recruitment process, participants were informed about the nature of the test, the length of time for results, and what procedures would be involved in self-administering the OQA test. After providing informed consent, including the release of information for research use, participants demonstrated their ability to properly take an OQA sample using a popsicle stick as a proxy for the testing device.
  Other Names: OraQuick Advance rapid test

SUMMARY:
The purpose of this study, conducted in Santiago-Chile, was to:

1. Evaluate the sensitivity and specificity of OraQuick Advance oral rapid test (OQA)when compared to ELISA;
2. Track the number of people in the study who returned for their ELISA test HIV results; and
3. Analyze the perception among participants of the use of OQA compared to ELISA testing for HIV screening.

DETAILED DESCRIPTION:
Human Immunodeficiency Virus /Acquired Immunodeficiency Syndrome (HIV/AIDS) continues to be one of the most devastating worldwide pandemics. In response to the HIV/AIDS epidemic, the Joint United Nations Programme on HIV/AIDS in 2010, urged countries to improve access to HIV/AIDS testing and counseling in an effort to increase the number of people who know their HIV status, thereby attempting to decrease transmission and increase treatment. Thus, an effective country response is to increase voluntary testing and counseling, particularly among at-risk populations. Ensuring patients receive their test results is an essential component of these efforts.

Chile, since 1991, has seen an increase of notified cases of HIV/ AIDS among certain regions of the country. The Chilean government offers free screening for HIV using only the ELISA test. In addition, many Chileans fail to return to receive their test results, as do many other individuals worldwide. In the United States, the Center for Disease Control reported that when using the "gold standard of HIV testing" (the ELISA) 30% of people with negative results and 39% of people with positive results do not return for their test results.

In Western counties, as well as several Latin American countries, the use of rapid testing technology to identify HIV 1 and 2 has increased the percentage of people who learn their serological status when compared with those who are tested using the traditional ELISA method. Neither the rapid test nor ELISA yield a definitive diagnosis, so further confirmation testing is required using the Western Blot to rule out the possibility of a false positive result. Nonetheless, by providing quick turn-around, rapid testing helps to facilitate individuals receiving their initial test results, thereby increasing the their probability of being quickly referred to appropriate health services for confirmatory testing and treatment.

Although the Food and Drug Administration (FDA) currently has approved six different rapid tests for clinical use to detect HIV 1 and 2, the OraQuick Advance Rapid Assessment (OQA) is the only one that is administered orally.

OQA testing can be conducted in geographical locations where laboratory facilities capable of performing ELISA assays are unavailable. Thus, HIV screening programs that adopt OQA can extend their reach far beyond previous locations.

Despite OQA's growing success and popularity in many different settings globally, Chile has yet to accept OQA or any rapid testing as a viable alternative to ELISA testing. The Chilean government has delayed approval for the adoption of OQA pending additional evidence among Chileans that it offers a more advantageous alternative to ELISA testing with equal specificity.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Seeking ELISA testing to learn their HIV status (group 1) or
* Having been confirmed HIV positive through Western Blot testing (Group 2)

Exclusion Criteria:

* HIV positive currently under antiretroviral medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 497 (Actual)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The sensitivity and specificity of a rapid test in oral fluid (OraQuick Advance)compare to the ELISA test for HIV. | 1 day (Immediately after the participants had taken their ELISA test for HIV or when recruited in case of people living with HIV.)
  OraQuick Advance rapid oral test (OQA) was administered to people living with HIV (PLWH) who were not under Anti-retroviral treatment. The PLWH had a previous positive ELISA test and confirmed diagnose with a Western-blot. People who didn't know their HIV diagnose, and who had come to the clinic for an ELISA test for HIV were also administered OQA test after they had completed their ELISA test.

SECONDARY OUTCOMES:
The number of people who received their result from the ELISA for HIV test, versus the number of people who receives their OQA results. | Clinic staff notified patient of their ELISA test results for up to three weeks after their clinic visit.
  Ones the results of the ELISA test came back from the laboratory, the responsible party at the clinic had to notify the patient and the research team about their ELISA for HIV result and if they had been successfully notifying the HIV status. The patient had authorized the clinic staff to disclosure their HIV result to the research team in the consent form when enrolled in the research. This results were compared with the number of people that would have received their result in the same visit (after 20 minutes) if administered OQA instead of the ELISA.

OTHER OUTCOMES:
Perceptions among study participants of the use of OQA compared to ELISA testing for HIV screening. | Within 3 months after they were administered their OQA test, the participants were either interviewed or participated in a focus group.
  Participants indicated their interest on their consent forms in being contacted at a later date to participate in a focus group or interview to discuss their testing experience and perceptions of both tests.

CONTACTS AND LOCATIONS:
Overall Officials: Lisette P Irarrazabal, PhD ©, Principal Investigator — Pontificia Universidad Catolica de Chile / University of Illinois at Chicago
Locations (1):
- School of Nursing, Pontificia Universidad Catolica de Chile, Macul, Santiago Metropolitan, Chile

REFERENCES:
- [Derived] Irarrazabal LP, Ferrer L, Cianelli R, Lara L, Reed R, Levy J, Perez C. Oral rapid test: an alternative to traditional HIV screening in Chile. Rev Panam Salud Publica. 2013 Jun;33(6):427-32. PMID 23939368